CLINICAL TRIAL: NCT02209896
Title: Safety and Performance of the BlueWind Medical Reprieve System for the Treatment of Patients With Peripheral Neuropathic Pain
Brief Title: BlueWind Reprieve System for the Treatment of PNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-04-001
Record Dates: First submitted 2014-08-03; First posted 2014-08-06 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Neuropathic Pain
Keywords: Peripheral Neuropathic Pain; PNP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BlueWind Reprieve System (Experimental): The Reprieve implant will be implanted for eligible patients. Implant parameters settings will be set according to patient's sensations.
  Interventions: Device: The Reprieve system

INTERVENTIONS:
Device: The Reprieve system — BlueWind Medical neurostimulator for the treatment of neuropathic pain

SUMMARY:
The BlueWind Reprieve system is a neurostimulator consisting of an Implant and external components.

The system is intended for home care use. The chronic pain treatment is achieved by an electrical stimulation of peripheral nerve fibers. The stimulation is set so that it generates paresthesia in the stimulated area (e.g. foot), reducing the pain sensation and improving the quality of life for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female aged 18 - 80.
* Patient agrees to attend all follow-up evaluations and is willing to completely and accurately fill out pain questionnaires.
* Diagnosis of chronic neuropathic pain due to peripheral neuropathy.
* Documented pain attributed to neuropathy for at least 6 months.
* Pain intensity with an average daily VAS score of at least 6, demonstrated by 3 ratings per day across 7 days.
* Patient refractory to conservative treatments including pain medication, for at least 6 months.
* Stable pain medication for at least 4 weeks prior to study enrollment.

Exclusion Criteria:

* Previous participation in another study with any investigational drug or device within the past 90 days.
* Any active implant (cardiac or other).
* Any metal implant in the area of BlueWind device implantation site.
* Current pregnancy or attempting to get pregnant (female patient).
* Any clinically significant neurologic disorders (except PNP).- Any clinically significant or unstable medical or psychiatric condition that would affect the patient's ability to participate in the study.
* Patients with severe or unstable cardiovascular, pulmonary, gastrointestinal, hematological, hepatic, renal or endocrine diseases.
* Severe peripheral vascular disease that may cause intermittent claudication or ischemic ulcers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The incidence of serious adverse events | 6 months
  The incidence of serious adverse events (system and/or procedure related events)
Pain assessment | 6 months post system activation
  Pain assessment by Visual Analogue Scale (VAS) as compared to baseline at 6 months post activation

SECONDARY OUTCOMES:
Clinical success defined as the effect of the Reprieve System on patient's symptoms | 6 months post system activation
  Measurements include:
  SF-McGill pain Questionnaire Pain related medication consumption/day Quality of life questionnaire SF-36 Health survey and safety

CONTACTS AND LOCATIONS:
Overall Officials: Ron Dabby, MD, Principal Investigator — Wolfson Medical Center
Locations (2):
- Israel (2):
  - Rambam Health care campus, Haifa
  - Edith Wolfson Medical Center, Holon